CLINICAL TRIAL: NCT00947856
Title: Treatment With SGN-35 in Patients With CD30-positive Hematologic Malignancies Who Have Previously Participated in an SGN-35 Study
Brief Title: A Brentuximab Vedotin Trial for Patients Who Have Previously Participated in a Brentuximab Vedotin Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-006; 2010-019932-11 (EudraCT Number)
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Drug Therapy; Hematologic Diseases; Immunotherapy; Monomethylauristatin E
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Hematologic Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BV Retreatment (Experimental): Brentuximab vedotin 1.2 or 1.8 mg/kg every 3 weeks by IV infusion (retreatment after relapse)
  Interventions: Drug: brentuximab vedotin
- BV Extension (Experimental): Brentuximab vedotin 1.2 or 1.8 mg/kg every 3 weeks by IV infusion (continued treatment)
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — Every 3 weeks by IV infusion (1.2 or 1.8 mg/kg) until disease progression, unacceptable toxicity, or study closure
  Other Names: Adcetris

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and efficacy of treatment with brentuximab vedotin (SGN-35) in patients who have previously participated in an brentuximab vedotin study.

DETAILED DESCRIPTION:
This is a multicenter, open-label study to evaluate single-agent brentuximab vedotin (SGN-35) treatment in patients who previously participated in a brentuximab vedotin study, including Studies SGN35-005 (NCT01100502), SGN35-007 (NCT01026233), and SGN35-008 (NCT01026415). Patients treated on this study (SGN35-006) could re-enroll on study if eligible. The study consisted of 2 arms, as follows:

* Retreatment arm: Patients with CD30-positive hematologic malignancies who experienced a complete remission (CR) or partial remission (PR) with previous brentuximab vedotin treatment on a clinical study and subsequently experienced disease progression or relapse. The purpose of this arm was to assess safety and efficacy of retreatment with brentuximab vedotin.
* Extension treatment arm: Patients with either CD30-positive hematologic or nonhematologic malignancies who completed treatment in a prior brentuximab vedotin study without unacceptable toxicity and experienced clinical benefit as assessed by the investigator. The purpose of this arm was to enable patients who participated in certain prior brentuximab vedotin trials to receive extension treatment and to assess patient safety and survival in the extension treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* Participated in a previous brentuximab vedotin study.
* CD30-positive hematologic malignancy.
* At a minimum, experienced clinical benefit in the prior brentuximab vedotin study. For retreatment, patients must have previously achieved either complete or partial remission with brentuximab vedotin and experienced disease progression after discontinuing the prior brentuximab vedotin study.

Exclusion Criteria:

Withdrew consent to participate in any prior brentuximab vedotin study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Grove, PA-C, Study Director — Seagen Inc.
Locations (17):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami Miller School of Medicine / Sylvester Comprehensive Cancer Center, Miami, Florida
  - Loyola University Medical Center - Cardinal Bernadin Cancer Center, Maywood, Illinois
  - St. Francis Medical Group Oncology & Hematology Specialists, Indianapolis, Indiana
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - The John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Clinical Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center /The University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance / University of Washington Medical Center, Seattle, Washington
- Hopital Saint-Louis/Service d'Hematologie, Paris, Cedex 10, France

REFERENCES:
- [Result] Bartlett NL, Chen R, Fanale MA, Brice P, Gopal A, Smith SE, Advani R, Matous JV, Ramchandren R, Rosenblatt JD, Huebner D, Levine P, Grove L, Forero-Torres A. Retreatment with brentuximab vedotin in patients with CD30-positive hematologic malignancies. J Hematol Oncol. 2014 Mar 19;7:24. doi: 10.1186/1756-8722-7-24. PMID 24642247
- [Derived] Gopal AK, Ramchandren R, O'Connor OA, Berryman RB, Advani RH, Chen R, Smith SE, Cooper M, Rothe A, Matous JV, Grove LE, Zain J. Safety and efficacy of brentuximab vedotin for Hodgkin lymphoma recurring after allogeneic stem cell transplantation. Blood. 2012 Jul 19;120(3):560-8. doi: 10.1182/blood-2011-12-397893. Epub 2012 Apr 17. PMID 22510871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Jul 2009 - Mar 2013
Period: Treatment Period
Arm/Group | BV Extension | BV Retreatment
Started | 78 | 32 (Two patients in extension arm re-enrolled in retreatment arm and are represented in both arms)
Completed | 0 | 0 (Patients treated until disease progression, unacceptable toxicity or study closure)
Not Completed | 78 | 32
Not completed — Progressive Disease | 33 | 12
Not completed — Adverse Event | 15 | 9
Not completed — Physician Decision | 14 | 6
Not completed — Study Stopped by Sponsor | 4 | 4
Not completed — Withdrawal by Subject | 12 | 1
Period: Follow-up Period
Arm/Group | BV Extension | BV Retreatment
Started | 78 | 32 (All participants were followed after treatment; thus, number started will not match number completed)
Completed | 27 | 9 (Completed survival follow-up due to death)
Not Completed | 51 | 23
Not completed — Study Stopped by Sponsor | 40 | 20
Not completed — Re-enrolled for Retreatment | 2 | 3
Not completed — Lost to Follow-up | 7 | 0
Not completed — Patient unavailable for site visits | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | BV Extension | BV Retreatment | Total
Number analyzed (Participants) | 78 | 32 | 110
Age, Customized [Median (Full Range); unit: years] | 32 [15 to 78] | 37 [16 to 72] | 33.5 [15 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 35 | 17 | 52
  Male | 43 | 15 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 4 | 11
  White | 66 | 27 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  France | 0 | 3 | 3
  United States | 78 | 29 | 107
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — 0 = Normal activity
  1. = Symptoms but ambulatory
  2. = In bed <50% of the time
  3. = In bed >50% of the time
  4. = 100% bedridden
  5. = Dead
  participants
    0 | 47 | 12 | 59
    1 | 30 | 18 | 48
    2 | 0 | 2 | 2
    3-5 | 0 | 0 | 0
    Missing | 1 | 0 | 1
Disease diagnosis [Number; unit: participants]
  Hodgkin lymphoma (HL) | 68 | 21 | 89
  Systemic anaplastic large cell lymphoma (ALCL) | 8 | 8 | 16
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate by Investigator
Description: Percentage of participants in the retreatment arm who achieved a best response of complete remission (CR, disappearance of all evidence of disease) or partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to approximately 38 months
Population: Any patient who received retreatment and had postbaseline response results; 1 HL patient did not have postbaseline response results and 3 ALCL patients were retreated more than once.
Measure: Number (95% Confidence Interval); unit: percentage of retreatment experiences
Units Other Than Participants: Retreatment Experiences
Groups:
- BV Retreatment - HL: Patients with Hodgkin lymphoma (HL) enrolled and treated on the retreatment arm
- BV Retreatment - ALCL: Patients with anaplastic large cell lymphoma (ALCL) enrolled and treated on the retreatment arm
- BV Retreatment - Other: Patients with other disease diagnoses enrolled and treated on the retreatment arm
- BV Retreatment Total: All patients enrolled and treated on the retreatment arm, including 3 patients retreated more than once
Arm/Group | BV Retreatment - HL | BV Retreatment - ALCL | BV Retreatment - Other | BV Retreatment Total
Number analyzed (Participants) | 21 | 8 | 3 | 32
Number analyzed (Retreatment Experiences) | 20 | 11 | 3 | 34
percentage of retreatment experiences | 60 [36.1 to 80.9] | 91 [58.7 to 99.8] | 33 [0.8 to 90.6] | 68 [49.5 to 82.6]

2. Primary Outcome: Adverse Events by Severity, Seriousness, and Relationship to Treatment
Description: Counts of participants who had adverse events or treatment-emergent adverse events (TEAE, defined as newly occurring or worsening after first dose on SGN35-006). Serious adverse events are reported from the time of informed consent. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 3.0) were used to assess severity (1=mild, 2=moderate, 3=severe, 4=life threatening/disabling, 5=death). Relatedness to study drug was assessed by the investigator (Yes/No). Participants with multiple occurrences of an adverse event within a category are counted once within the category.
Time Frame: up to 39 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | BV Extension | BV Retreatment
Number analyzed (Participants) | 78 | 32
participants
  Any TEAE | 75 | 31
  TEAE related to study drug | 65 | 27
  TEAE with severity grade >/=3 | 37 | 16
  Discontinued treatment due to adverse event | 13 | 9
  Serious adverse event | 16 | 9
  Serious adverse event related to study drug | 10 | 4

3. Primary Outcome: Laboratory Abnormalities >/= Grade 3
Description: Counts of study participants with post-baseline laboratory abnormalities of Grade 3 or greater per NCI CTCAE version 3.0. Participants with multiple occurrences of a laboratory abnormality within a category are counted once in that category.
Time Frame: Up to 39 months
Population: All participants who received treatment
Measure: Number; unit: participants
Arm/Group | BV Extension | BV Retreatment
Number analyzed (Participants) | 78 | 32
participants
  Any >/= Grade 3 laboratory abnormality | 29 | 12
  Lymphocytes (low) | 16 | 8
  Leukocytes (low) | 3 | 3
  Neutrophils (low) | 7 | 3
  Phosphate (low) | 7 | 3
  Platelets (low) | 4 | 3
  Aspartate aminotransferase (high) | 1 | 2
  Glucose (high) | 3 | 2
  Alanine aminotransferase (high) | 1 | 1
  Bilirubin (high) | 0 | 1
  Calcium (low) | 0 | 1
  Hemoglobin (low) | 1 | 1
  Potassium (low) | 0 | 1
  Sodium (low) | 2 | 0

4. Secondary Outcome: Duration of Objective Response by Kaplan-Meier Analysis
Description: Duration of objective response (CR + PR) on retreatment, defined as time of initial response until disease progression or death
Time Frame: Up to 38 months
Population: Participants with objective response among those who received retreatment
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Retreatment Experiences
Arm/Group | BV Retreatment - HL | BV Retreatment - ALCL | BV Retreatment - Other | BV Retreatment Total
Number analyzed (Participants) | 21 | 8 | 3 | 32
Number analyzed (Retreatment Experiences) | 12 | 10 | 1 | 23
months | 9.2 [2.1 to NA] — Insufficient number of events to estimate upper bound | 8.8 [1.4 to 12.9] | NA [NA to NA] — Insufficient number of events to estimate median and upper and lower bounds | 9.2 [6.6 to 12.9]

5. Secondary Outcome: Progression-free Survival by Kaplan-Meier Analysis
Description: Progression-free survival, defined as time from start of study treatment in the retreatment arm to disease progression per investigator or death due to any cause
Time Frame: Up to approximately 29 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Retreatment Experiences
Arm/Group | BV Retreatment - HL | BV Retreatment - ALCL | BV Retreatment - Other | BV Retreatment Total
Number analyzed (Participants) | 21 | 8 | 3 | 32
Number analyzed (Retreatment Experiences) | 20 | 11 | 3 | 34
months | 9.9 [3.4 to 13.4] | 12.9 [3.4 to 18.5] | 4.4 [1.2 to NA] — Insufficient number of events to estimate upper bound | 9.9 [4.4 to 13.4]

6. Secondary Outcome: Overall Survival
Description: Overall survival for both extension and retreatment arms, defined as time from start of study treatment to date of death due to any cause
Time Frame: Up to approximately 41 months
Population: Patients who received treatment on the extension arm, and patients who received retreatment and had postbaseline response results; 1 HL patient on the retreatment arm did not have postbaseline response results and 3 ALCL patients on the retreatment arm were retreated more than once.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Retreatment or Extension Trt Experiences
Groups:
- BV Extension Total: All patients enrolled and treated on the extension arm
Arm/Group | BV Extension Total | BV Retreatment - HL | BV Retreatment - ALCL | BV Retreatment - Other | BV Retreatment Total
Number analyzed (Participants) | 78 | 21 | 8 | 3 | 32
Number analyzed (Retreatment or Extension Trt Experiences) | 78 | 20 | 11 | 3 | 34
months | NA [32.1 to NA] — Insufficient number of events to estimate median and upper bound | NA [11.4 to NA] — Insufficient number of events to estimate median and upper bound | NA [NA to NA] — Insufficient number of events to estimate median and upper and lower bounds | NA [5.1 to NA] — Insufficient number of events to estimate median and upper bound | NA [19.5 to NA] — Insufficient number of events to estimate median and upper bound

7. Secondary Outcome: Incidence of Antitherapeutic Antibodies
Description: Counts of participants with anti-brentuximab vedotin antibodies at any time during extension treatment on Study SGN35-006 or number of retreatment experiences with anti-brentuximab vedotin antibodies at any time during retreatment
Time Frame: Up to 39 months
Population: Any patient who received extension treatment or retreatment and had baseline and postbaseline sample results; 1 HL patient on the retreatment arm did not have postbaseline sample results and 3 ALCL patients on the retreatment arm were retreated more than once and had samples.
Measure: Number; unit: participants or experiences
Units Other Than Participants: Retreatment or Extension Txt Experiences
Arm/Group | BV Extension | BV Retreatment
Number analyzed (Participants) | 78 | 31
Number analyzed (Retreatment or Extension Txt Experiences) | 78 | 34
participants or experiences | 15 | 12

ADVERSE EVENTS:
Description: Treatment-emergent adverse events (TEAEs) defined as newly occurring (not present at baseline) or worsening after first dose of investigational product on Study SGN35-006
Groups:
- BV Extension; BV Retreatment: Brentuximab vedotin 1.2 or 1.8 mg/kg every 3 weeks by IV infusion
Arm/Group | BV Extension | BV Retreatment
Serious Adverse Events (participants affected / at risk) | 16/78 | 9/32
Other Adverse Events (participants affected / at risk) | 75/78 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BV Extension (N=78) | BV Retreatment (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Necrotising retinitis (Eye disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Graft versus host disease (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Small intestine obstruction (Gastrointestinal disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BV Extension (N=78) | BV Retreatment (N=32)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Neutropenia (Blood and lymphatic system disorders) | 10 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Tachycardia (Cardiac disorders) | 4 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 12
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 19 | 12
Chills (General disorders) | 5 | 2
Fatigue (General disorders) | 23 | 11
Infusion site extravasation (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 6 | 4
Oedema peripheral (General disorders) | 7 | 5
Pyrexia (General disorders) | 20 | 8
Hypogammaglobulinaemia (Immune system disorders) | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 25 | 6
Urinary tract infection (Infections and infestations) | 0 | 3
Skin injury (Injury, poisoning and procedural complications) | 0 | 3
Weight decreased (Investigations) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 11 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 3
Dizziness (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 10 | 9
Paraesthesia (Nervous system disorders) | 4 | 2
Peripheral motor neuropathy (Nervous system disorders) | 4 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 36 | 17
Syncope (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 4 | 3
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Flushing (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 12 | 0
Chest discomfort (General disorders) | 4 | 0
Pain (General disorders) | 6 | 0
Herpes zoster (Infections and infestations) | 7 | 0
Pneumonia (Infections and infestations) | 5 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.